CLINICAL TRIAL: NCT05026502
Title: Real-world Experience of Elagolix With E2/NETA for the Treatment of Heavy Menstrual Bleeding (HMB) Associated With Uterine Fibroids (UF): an Observational Study (The REACH Study)
Brief Title: A Study to Assess Patient-Reported Quality of Life and Effectiveness on Control of Bleeding in Adult Participants With Heavy Menstrual Bleeding Due to Uterine Fibroids Taking Oral Oriahnn Capsules
Acronym: REACH
Status: Terminated | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-296
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Heavy Menstrual Bleeding; Uterine Fibroids
Keywords: Elagolix; Estradiol/Norethindrone Acetate (E2/NETA); Oriahnn; ABT-620; Heavy Menstrual Bleeding (HMB); Uterine Fibroids (UF)
MeSH Terms: conditions — Menorrhagia; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Being Treated With Elagolix + E2/NETA: Participants will receive Elagolix with Estradiol/Norethindrone Acetate per Standard of Care, as prescribed by their physicians.

SUMMARY:
Uterine Fibroids (UF) are noncancerous (benign) tumors that commonly occur in up to 80% of women of reproductive age. Symptoms can include heavy menstrual bleeding (HMB), low back pain, urinary frequency and urgency, gastrointestinal symptoms, and fatigue. In participants with UF, this study will prospectively assess changes in patient-reported quality of life and patient-reported effectiveness in controlling HMB when treated with elagolix, estradiol, and norethindrone acetate capsules; elagolix capsules (elagolix + E2/NETA).

Around 200 adult premenopausal female participants in the United States with a diagnosis of HMB associated with UF and are prescribed elagolix + E2/NETA by their physicians as per standard of care will be enrolled in this direct-to-patient observational study for up to 6 months.

Participants will have been prescribed elagolix + E2/NETA within the last 30 days prior to enrollment and will continue to take elagolix + E2/NETA throughout study participation.

There may be a higher burden for participants in this study compared to standard of care. Electronic patient reported outcomes (ePROs) will be collected at baseline, 1, 3 and 6 months to assess the impact of Elagolix + E2/NETA on patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have initiated elagolix + Estradiol/Norethindrone Acetate (E2/NETA) in the last 30 days or less, or with planned initiation of elagolix + E2/NETA prescribed as part of standard of care treatment.
* Participants self-reporting heavy menstrual bleeding (HMB) associated with uterine fibroids (UF).
* Participants are premenopausal (i.e., still report experiencing menses).

Exclusion Criteria:

* Participants that report they are pregnant or planning to become pregnant in next 6 months.
* Participants reporting a surgical history of:

  * Hysterectomy (with or without oophorectomy).
  * Bilateral oophorectomy.
* Participants who have initiated elagolix + E2/NETA more than 30 days ago.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult female participants diagnosed with heavy menstrual bleeding associated with uterine fibroids who have been prescribed elagolix + E2/NETA as part of standard of care
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Self-Reported Heavy Menstrual Bleeding (HMB) Measured by Menstrual Bleeding Questionnaire (MBQ) | Up to 3 Months
  MBQ is a self-reported questionnaire that measures impact of HMB with 20 items and includes perception of heaviness of bleeding, bleeding pattern, pain, and impact of symptoms including social embarrassment, fear of social embarrassment, and behavioral changes to avoid social embarrassment. Sum responses to obtain a total score and multiply score by 1.32 to scale. Zero, least impact possible; 100, worst impact possible.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- IQVIA RDS, Inc., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-296#additional-resources-section